CLINICAL TRIAL: NCT02540902
Title: A Prospective Study of an All Polyethylene Tibial Component Used in Total Knee Arthroplasty Surgery
Brief Title: Study of an All Polyethylene Tibial Component
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Golden Jubilee National Hospital (Other Government)
Collaborators: Aesculap AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Ortho 15-06
Record Dates: First submitted 2015-08-11; First posted 2015-09-04 (Estimated); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Knee Replacement
Keywords: Knee replacement; Knee arthroplasty; All-polyethylene tibia; Bone density

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All-poly (Experimental): Knee arthroplasty with all-polyethylene tibia
  Interventions: Device: All-polyethylene tibia (Aesculap AG)

INTERVENTIONS:
Device: All-polyethylene tibia (Aesculap AG) — Implantation of an all polyethylene tibial component.
  Other Names: Aesculap All Poly Tibia Plateau Columbus CR DD; NN1200-NN1203, NN1210-NN1213, NN1220-NN1223; NN1230-NN1233, NN1240-NN1243, NN1250-NN1253

SUMMARY:
This will be a prospective single cohort investigation of the Columbus all polyethylene tibia (Aesculap AG, Tuttlingen, Germany) used in total knee arthroplasty (TKA) surgery. The aim of the project is to determine post-operative outcome of the all polyethylene tibia up to two years.

DETAILED DESCRIPTION:
Thirty consecutive TKA patients under the care of two orthopaedic consultants at the Golden Jubilee National Hospital who meet the inclusion/exclusion criteria will be recruited to the study and will be given the all polyethylene tibia. Participants will return for their standard postoperative followup appointments (6 weeks and 1 year post-operatively). In addition to standard care, a bone density scan using dual energy x-ray absorptiometery (DXA) will be done as part of the 6 weeks post-operative follow-up. A second DXA scan will be done at an additional appointment at the hospital between 18 and 24 months post-operatively for a bone density scan which is not part of standard care.

The data which will be analysed will be the results of the bone scan, computer generated data about the range of movement (RoM) and alignment of the operated knee collected as part of the operation, the RoM, clinical outcome and satisfaction data collected at the pre-operative assessment and post-operative followups, pre- and post-operative x-rays, complications, survivorship and surgeon experience of using the all polyethylene tibia. These data will be investigated to see if the all polyethylene tibia has satisfactory outcomes with no adverse effects.

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral TKA
2. Aged 70 year or older
3. BMI < 37.5
4. Suitable to receive the study implant

Exclusion Criteria:

1. Revision of existing knee replacement
2. Previous lower limb replacement
3. Proximal tibial bone defects
4. Diagnosed osteopenia or osteoporosis
5. Unable to give informed consent
6. Unwilling to take part
7. Unable to return to the Golden Jubilee National Hospital for followup appointments

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density | 18 to 24 months post-operatively
  Measure of peri-prosthetic bone mineral density

SECONDARY OUTCOMES:
Intra-operative RoM | Intra-operative
  Range of movement of the knee joint measured by the navigation computer during surgery
Intra-operative alignment | Intra-operative
  The leg alignment measured by the navigation computer during surgery.
RoM | 1 year
  Active range of motion of the knee joint
Oxford Knee Score | 1 year
  Clinical outcome measure
EQ-5D | 1 year
  General health measure
Patient satisfaction | 1 year
  Patient satisfaction with surgery (Scale: 0 to 10, 0 = not satisfied, 10 = very satisfied)
Leg alignment | 1 year
  Leg alignment measured from long leg x-rays
Bone condition | 1 year
  Signs of osteolysis from knee x-rays
Complications | 1 year
  Any post-operative complications as a result of surgery, e.g. infection, revision, aseptic loosening.
Implant survivorship | 18 to 24 months
  Percentage of implants still in situ over time.
Surgeon feedback from surgery | intra-operative
  Surgeon experience and issues with using all-polyethylene tibia using an un-validated questionnaire.
Component position | 1 year
  Migration of the component over time measured from x-rays
Peri-prosthetic lucency | 1 year
  Radiolucent lines (>2mm wide) around the component which may indicate component loosening

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Picard, MD, Principal Investigator — Golden Jubilee National Hospital
Locations (1):
- Golden Jubilee National Hospital, Clydebank, West Dunbartonshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No